CLINICAL TRIAL: NCT03572257
Title: Prospective, Double-Blind, Randomized Controlled Trial of Quetiapine as a Treatment for Delirium in Critically Ill Children
Brief Title: Quetiapine Treatment for Pediatric Delirium
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Closed due to inability to enroll
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Rita Alvarez, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1195004
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Quetiapine (0.5 mg/kg TID x 10 days) (Experimental): This study group will receive treatment with quetiapine after diagnosis of pediatric delirium. Group assignment will be blinded.
  Interventions: Drug: Quetiapine
- Placebo (Placebo Comparator): This study group will receive a placebo treatment after diagnosis of pediatric delirium. Group assignment will be blinded.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Quetiapine — Patients randomized to the study treatment group will received quetiapine at 0.5 mg/kg, three times a day for 10 days. Doses can be increased up to a maximum of 6 mg/kg/day, in increments of 0.5 mg/kg, based on the subject's clinical delirium symptoms. PRN doses of 0.5 mg/kg can be given up to three times a day based on the clinical judgement of the subject's ICU care team.
  Arms: Quetiapine (0.5 mg/kg TID x 10 days)
Other: Placebo — Patients randomized to the placebo group will be given an equivalent volume of sterile liquid or sugar pill, based on the individual subjects dosing preference or ability. Dosing will be done on the same schedule as the quetiapine group
  Arms: Placebo

SUMMARY:
This is a prospective, double-blind, randomized controlled trial to begin determining the efficacy of quetiapine as a treatment for pediatric delirium in patients admitted to the pediatric intensive care unit (PICU)

DETAILED DESCRIPTION:
Delirium is an acute syndrome with fluctuation in mental status with altered cognition and consciousness. It is a common occurrence (17% to 38%) in critically ill children with serious short-term consequences. Its pathophysiology is complex and incompletely understood. Dopaminergic, serotoninergic, glutaminergic, and cholinergic pathways in the cerebral cortex, striatum, substantia nigra, and thalamus have been implicated. Imbalance in the synthesis, release, and inactivation of neurotransmitters can result in altered cognitive function, behavior, and mood. The Society of Critical Care Medicine set the adult practice guidelines including widespread delirium screening as well as treatment to decrease duration of delirium and ameliorate its long-term effects (12). The cornerstone of pharmacologic therapy for delirium in adults is antipsychotics, both first and second-generation (13-20).

The current foundation of treatment for pediatric delirium is identifying and addressing the underlying etiology. Iatrogenic factors should be minimized, such as avoiding benzodiazepines and restraints, optimizing pain control, minimizing sedation, and treating withdrawal. The ICU environment should also be optimized to create a quiet, well-lit space with clustered care to allow for uninterrupted sleep. When non-pharmacologic treatment measures prove insufficient to manage the symptoms of delirium, we believe the second-generation antipsychotic (SGA) quetiapine may have a role in the treatment of delirium. However, there are currently no FDA-approved medications to treat delirium in this population.

The European Society of Paediatric and Neonatal Intensive Care (ESPNIC) has recently recommended that all children in the ICU be monitored for delirium but provided no guidance on recommended treatments (21), likely due to the lack of evidence of proven delirium treatment in children. An adult systematic review and meta-analysis by Kishi et al concluded that antipsychotics are superior to placebo in decreasing severity of delirium and time to response with there was no significant difference in the side effects between the two groups. Additionally, SGAs are associated with a shorter time to response and lower side effect profile than haloperidol (a first-generation antipsychotic).

A growing body of pediatric literature suggests that delirium is a serious and under recognized problem in critically ill children as well, however little research has been focused on treatment . A recent retrospective series looking at the use of quetiapine in suggested that quetiapine use for delirium treatment is a safe option in this population.

With proven efficacy in adults with delirium, an established track record in children for indications other than delirium, a favorable safety profile, and a wide therapeutic window, quetiapine is a logical choice for the next phase of research into pediatric delirium treatment. In this study are looking prospectively at the effectiveness of quetiapine as a treatment for pediatric delirium.

ELIGIBILITY:
Inclusion Criteria:

* Age 0 - 21 years old
* PICU admission
* Positive CAPD scoring

  * For developmentally normal children a CAPD score of ≥ 9
  * For developmentally delayed a CAPD score of ≥ 9 and a Richmond Agitation Sedation Scale (RASS) fluctuation of at least 2 points in the last 24 hours

Exclusion Criteria:

* Patients under neuromuscular blockade and/or therapeutic hypothermia.
* Patients undergoing treatment of alcohol withdrawal.
* Patients unable to tolerate enteral medications
* Patients on antipsychotics
* Patients with a history of:

  * hepatic encephalopathy, hepatitis
  * elevated liver enzymes defined ALT or AST above normal range for age since hospitalization
  * baseline QTc prolongation (defined as greater than 97th percentile for age or greater than 20% increase from baseline or previous QTc)
  * major depressive disorder or bipolar disorder, and movement disorder.
* Patients who are pregnant
* Non-English and non-Spanish speaking subjects and/or parent/guardian

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Time to resolution of delirium | Screening through Study Day 14/Hospital Discharge
  Delirium symptoms will be monitored using CAPD (Cornell Assessment for Pediatric Delirium) score, collected twice a day. Time to resolution of delirium will be measured from the time of randomization to the time scores are within normal range (0-8). Number of days with abnormal CAPD scores will be compared between study groups

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Traube C, Silver G, Reeder RW, Doyle H, Hegel E, Wolfe HA, Schneller C, Chung MG, Dervan LA, DiGennaro JL, Buttram SD, Kudchadkar SR, Madden K, Hartman ME, deAlmeida ML, Walson K, Ista E, Baarslag MA, Salonia R, Beca J, Long D, Kawai Y, Cheifetz IM, Gelvez J, Truemper EJ, Smith RL, Peters ME, O'Meara AM, Murphy S, Bokhary A, Greenwald BM, Bell MJ. Delirium in Critically Ill Children: An International Point Prevalence Study. Crit Care Med. 2017 Apr;45(4):584-590. doi: 10.1097/CCM.0000000000002250. PMID 28079605
- [Background] Traube C, Silver G, Gerber LM, Kaur S, Mauer EA, Kerson A, Joyce C, Greenwald BM. Delirium and Mortality in Critically Ill Children: Epidemiology and Outcomes of Pediatric Delirium. Crit Care Med. 2017 May;45(5):891-898. doi: 10.1097/CCM.0000000000002324. PMID 28288026
- [Background] Traube C, Greenwald BM. "The Times They Are A-Changin": Universal Delirium Screening in Pediatric Critical Care. Pediatr Crit Care Med. 2017 Jun;18(6):594-595. doi: 10.1097/PCC.0000000000001142. No abstract available. PMID 28574907
- [Background] Schieveld JN, Strik JJ. Pediatric Delirium: A Worldwide PICU Problem. Crit Care Med. 2017 Apr;45(4):746-747. doi: 10.1097/CCM.0000000000002275. No abstract available. PMID 28291099
- [Background] Patel AK, Biagas KV, Clarke EC, Gerber LM, Mauer E, Silver G, Chai P, Corda R, Traube C. Delirium in Children After Cardiac Bypass Surgery. Pediatr Crit Care Med. 2017 Feb;18(2):165-171. doi: 10.1097/PCC.0000000000001032. PMID 27977539
- [Background] Meyburg J, Dill ML, Traube C, Silver G, von Haken R. Patterns of Postoperative Delirium in Children. Pediatr Crit Care Med. 2017 Feb;18(2):128-133. doi: 10.1097/PCC.0000000000000993. PMID 27776085
- [Background] Leroy PL, Schieveld JN. Mind the Heart: Delirium in Children Following Cardiac Surgery for Congenital Heart Disease. Pediatr Crit Care Med. 2017 Feb;18(2):196-198. doi: 10.1097/PCC.0000000000001038. No abstract available. PMID 28157798
- [Background] Traube C, Mauer EA, Gerber LM, Kaur S, Joyce C, Kerson A, Carlo C, Notterman D, Worgall S, Silver G, Greenwald BM. Cost Associated With Pediatric Delirium in the ICU. Crit Care Med. 2016 Dec;44(12):e1175-e1179. doi: 10.1097/CCM.0000000000002004. PMID 27518377
- [Background] Smith HA, Gangopadhyay M, Goben CM, Jacobowski NL, Chestnut MH, Savage S, Rutherford MT, Denton D, Thompson JL, Chandrasekhar R, Acton M, Newman J, Noori HP, Terrell MK, Williams SR, Griffith K, Cooper TJ, Ely EW, Fuchs DC, Pandharipande PP. The Preschool Confusion Assessment Method for the ICU: Valid and Reliable Delirium Monitoring for Critically Ill Infants and Children. Crit Care Med. 2016 Mar;44(3):592-600. doi: 10.1097/CCM.0000000000001428. PMID 26565631
- [Background] Porter S, Holly C, Echevarria M. Infants with Delirium: A Primer on Prevention, Recognition, and Management. Pediatr Nurs. 2016 Sep-Oct;42(5):223-9. PMID 29406640
- [Background] Maldonado JR. Neuropathogenesis of delirium: review of current etiologic theories and common pathways. Am J Geriatr Psychiatry. 2013 Dec;21(12):1190-222. doi: 10.1016/j.jagp.2013.09.005. PMID 24206937
- [Background] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med. 2013 Jan;41(1):263-306. doi: 10.1097/CCM.0b013e3182783b72. PMID 23269131
- [Background] Kishi T, Hirota T, Matsunaga S, Iwata N. Antipsychotic medications for the treatment of delirium: a systematic review and meta-analysis of randomised controlled trials. J Neurol Neurosurg Psychiatry. 2016 Jul;87(7):767-74. doi: 10.1136/jnnp-2015-311049. Epub 2015 Sep 4. PMID 26341326
- [Background] Bathula M, Gonzales JP. The pharmacologic treatment of intensive care unit delirium: a systematic review. Ann Pharmacother. 2013 Sep;47(9):1168-74. doi: 10.1177/1060028013500466. PMID 24259732
- [Background] Boettger S, Friedlander M, Breitbart W, Passik S. Aripiprazole and haloperidol in the treatment of delirium. Aust N Z J Psychiatry. 2011 Jun;45(6):477-82. doi: 10.3109/00048674.2011.543411. PMID 21563866
- [Background] Banerjee A, Girard TD, Pandharipande P. The complex interplay between delirium, sedation, and early mobility during critical illness: applications in the trauma unit. Curr Opin Anaesthesiol. 2011 Apr;24(2):195-201. doi: 10.1097/ACO.0b013e3283445382. PMID 21386669
- [Background] Martin J, Heymann A, Basell K, Baron R, Biniek R, Burkle H, Dall P, Dictus C, Eggers V, Eichler I, Engelmann L, Garten L, Hartl W, Haase U, Huth R, Kessler P, Kleinschmidt S, Koppert W, Kretz FJ, Laubenthal H, Marggraf G, Meiser A, Neugebauer E, Neuhaus U, Putensen C, Quintel M, Reske A, Roth B, Scholz J, Schroder S, Schreiter D, Schuttler J, Schwarzmann G, Stingele R, Tonner P, Trankle P, Treede RD, Trupkovic T, Tryba M, Wappler F, Waydhas C, Spies C. Evidence and consensus-based German guidelines for the management of analgesia, sedation and delirium in intensive care--short version. Ger Med Sci. 2010 Feb 2;8:Doc02. doi: 10.3205/000091. PMID 20200655
- [Background] Straker DA, Shapiro PA, Muskin PR. Aripiprazole in the treatment of delirium. Psychosomatics. 2006 Sep-Oct;47(5):385-91. doi: 10.1176/appi.psy.47.5.385. PMID 16959926
- [Background] Boettger S, Breitbart W. Atypical antipsychotics in the management of delirium: a review of the empirical literature. Palliat Support Care. 2005 Sep;3(3):227-37. doi: 10.1017/s1478951505050352. PMID 16594462
- [Background] Ely EW, Stephens RK, Jackson JC, Thomason JW, Truman B, Gordon S, Dittus RS, Bernard GR. Current opinions regarding the importance, diagnosis, and management of delirium in the intensive care unit: a survey of 912 healthcare professionals. Crit Care Med. 2004 Jan;32(1):106-12. doi: 10.1097/01.CCM.0000098033.94737.84. PMID 14707567
- [Background] Harris J, Ramelet AS, van Dijk M, Pokorna P, Wielenga J, Tume L, Tibboel D, Ista E. Clinical recommendations for pain, sedation, withdrawal and delirium assessment in critically ill infants and children: an ESPNIC position statement for healthcare professionals. Intensive Care Med. 2016 Jun;42(6):972-86. doi: 10.1007/s00134-016-4344-1. Epub 2016 Apr 15. PMID 27084344
- [Background] Devlin JW, Roberts RJ, Fong JJ, Skrobik Y, Riker RR, Hill NS, Robbins T, Garpestad E. Efficacy and safety of quetiapine in critically ill patients with delirium: a prospective, multicenter, randomized, double-blind, placebo-controlled pilot study. Crit Care Med. 2010 Feb;38(2):419-27. doi: 10.1097/CCM.0b013e3181b9e302. PMID 19915454
- [Background] Joyce C, Witcher R, Herrup E, Kaur S, Mendez-Rico E, Silver G, Greenwald BM, Traube C. Evaluation of the Safety of Quetiapine in Treating Delirium in Critically Ill Children: A Retrospective Review. J Child Adolesc Psychopharmacol. 2015 Nov;25(9):666-70. doi: 10.1089/cap.2015.0093. Epub 2015 Oct 15. PMID 26469214